CLINICAL TRIAL: NCT05297955
Title: A Retrospective Study of Data Related to Circulating Tumor Cell Detection in Hepatocellular Carcinoma
Brief Title: Circulating Tumor Cell Detection in Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaoping, Chair of surgery department, Tongji Hospital
Other Study IDs: TJ-IRB20211242
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Circulating Tumor Cell
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The number of CTC in HCC patient great than or equal to two: According to the cutoff of CTC, the number of CTC in HCC patient great than or equal to two
- The number of CTC in HCC patient less than two: According to the cutoff of CTC,the number of CTC in HCC patient less than two

SUMMARY:
The investigators examined circulating tumor cells (CTC) in the perioperative peripheral blood of hundreds of HCC patients undergoing liver cancer surgery using CellSearch technology between 2013 and 2016. Although the investigators have done a preliminary study of the above data and published some results, the previous study was only a basic analysis. Now the investigators plan to carry out further in-depth analysis of these data, including hospitalization data, follow-up results, surgical tumors and blood specimens, and make full use of biostatistics, molecular biology, pathology and other related techniques to elucidate the association between the levels of CTC or CTC clusters and patients' disease during the perioperative period, and to explore the molecular basis of CTC production in hepatocellular carcinoma.

DETAILED DESCRIPTION:
From 2013 to 2016, CellSearch technology was used to detect the number of circulating tumor cells (CTC) in peripheral blood of hundreds of HCC patients undergoing liver cancer surgery during perioperative period. The analysis results confirmed that the level of CTC before and after surgery were significantly correlated with overall survival (OS) and disease-free survival (DFS) of patients. CTC level changed before and after surgery, but there was no statistical difference. Preoperative CTC was more correlated with patients' disease-related clinical parameters, while postoperative CTC was an independent prognostic indicator of patients after surgery. In addition, the investigators' study found that CTC clusters level can be a new marker of tumor progression in HCC patients.

Based on the above data, the investigators will perform retrospective analysis to compare the relationship between CTC level and clinical indicators of HCC patients. Participants were divided into groups according to pathological type, differentiation degree, clinical stage, invasion degree, recurrence and metastasis of tumors. Combined with immunohistochemistry and quantitative PCR results, the correlation of CTC in tumor genesis, pathological model, degree of differentiation, tumor stage, invasion, metastasis and expression of other tumor markers was studied.

ELIGIBILITY:
Inclusion Criteria:

* The pathological diagnosis was primary liver cancer.
* Undergoing radical surgical treatment
* No preoperative antitumor therapy was received
* Between 18 and 80 years old

Exclusion Criteria:

* With distal metastasis
* With other tumors
* Perioperative death
* Recurrence within one month after surgery
* Lost contact before the first follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Perioperative patients with hepatocellular carcinoma who underwent CTC detection of peripheral blood
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Data analysis of relationship between CTC and pathological indicators of hepatocellular carcinoma | 2022.03.15
  The previous CTC detection data of 458 cases was collected. To compare the relationship between CTC level of perioperative peripheral blood and clinical indexes of HCC patients, the main statistical analysis were one-way ANOVA, Student's T test and Multivariable Cox regression.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No